CLINICAL TRIAL: NCT05572710
Title: Avalus European Registry - an Observational Study to Evaluate Safety and Efficacy in a Real World Population
Acronym: Avalus
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S63824
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, observational, single-arm, multi-center registry of patients undergoing bioprosthetic aortic valve replacement with the Avalus valve. This prospective registry aims to examine the outcome and performance of surgical aortic valve replacement with the Avalus pericardial bioprosthesis.

DETAILED DESCRIPTION:
The study is a prospective, observational, single-arm, multi-center registry. The patients must undergoing bioprosthetic aortic valve replacement with the Avalus valve. This prospective registry aims to examine the outcome and performance of surgical aortic valve replacement with the Avalus pericardial bioprosthesis.

The goal of this project is to evaluate the real world results of aortic valve replacement with the Avalus valve. This will result in clinical and hemodynamic knowledge of this particular valve. The investigators are aiming for 1000 patient inclusions distributed over 40 sites across Europe and potentially also involving Canada.

Intentionally, we kept the inclusion criteria as wide as possible in order to obtain a real-world experience with and performance of the bioprosthesis. Patients younger than 18 years and salvage procedures are the only exclusion criteria from the registry. Outcome is evaluated in accordance with the VARC-2 criteria up to 1-year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for replacement of the native or prosthetic aortic valve with a bioprosthesis
* Age >= 18 years
* Patient has been adequately informed of risks and requirements of the registry (which are actually limited since the prosthesis is in full commercial use and only data registration is performed) and is able to provide informed consent for participation in the clinical registry.

Exclusion Criteria:

* Patient requires salvage surgery (according to EuroSCORE II definitions: "patients requiring cardiopulmonary resuscitation (external cardiac massage) en route to the operating theatre or prior to induction of anaesthesia. This does not include cardiopulmonary resuscitation following induction of anaesthesia")
* Not been able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real world population indicated for aortic valve replacement
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality and disabling stroke | 1 year
  Composite of all-cause mortality and disabling stroke

SECONDARY OUTCOMES:
VARC-2 | 1 year
  Mortality, stroke, bleeding complications, major vascular complications, new pacemaker implantation, prostethic valve function, composit endpoints

CONTACTS AND LOCATIONS:
Locations (19):
- Belgium (5):
  - UZ Leuven, Leuven, Vlaams-Brabant
  - UCL St Luc, Brussels
  - ZOL, Genk
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
- Rigshospitalet, Copenhagen, Denmark
- Kuopio University Hospital, Kuopio, Finland
- CHU Nantes, Nantes, France
- Germany (2):
  - Schüchtermann-Klinik, Bad Rothenfelde
  - Universität Herzzentrum, Hamburg
- Italy (6):
  - Osp. S.Orsola Malpighi, Bologna
  - Fondazione Poliambulanza, Brescia
  - Villa Maria Cecilia, Cotignola
  - Policlinico San Donato S.P.A, Milan
  - European Hospital, Roma
  - A. Sanitaria O. Ordine Mauriziano, Torino
- UMC Maastricht, Maastricht, Netherlands
- Spain (2):
  - Hospital Rambla, Santa Cruz de Tenerife
  - Hospital Clinico De Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No